CLINICAL TRIAL: NCT02987868
Title: Effects of an Amino Acid-Based hGH Secretagogue on Triiodythyronine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PBRC 10043 - HGH/Somatostatin
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Growth Hormone Treatment; Aging
Keywords: Somatostatin; Thyroid Hormone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement 1st day, placebo 2nd day (Active Comparator): Administration of oral supplement (proprietary amino acid derivative blend). Half of the participants took the Amino acid supplement first day and half of the participants took the Amino acid supplement second day.
  Interventions: Drug: Amino acid supplement first day; Drug: Placebo second day
- Placebo 1st day, supplement 2nd day (Placebo Comparator): Half of the participants took the placebo first day and half of the participants took placebo second day.
  Interventions: Drug: Placebo first day; Drug: Amino acid supplement second day

INTERVENTIONS:
Drug: Amino acid supplement first day — An orally administered supplement of the proprietary amino acid derivative
  Other Names: SeroVital™
  Arms: Supplement 1st day, placebo 2nd day
Drug: Placebo first day — A non-active orally administered supplement of the proprietary amino acid derivative
  Other Names: Non-active
  Arms: Placebo 1st day, supplement 2nd day
Drug: Amino acid supplement second day — An orally administered supplement of the proprietary amino acid derivative
  Other Names: SeroVital™
  Arms: Placebo 1st day, supplement 2nd day
Drug: Placebo second day — A non-active orally administered supplement of the proprietary amino acid derivative
  Other Names: Non-active
  Arms: Supplement 1st day, placebo 2nd day

SUMMARY:
In a recent randomized, double-blind, cross-over clinical trial, serum growth hormone (hGH) increased 682% above baseline 120 minutes after oral administration of an amino acid-based dietary supplement (SeroVital), p=0.01 vs placebo. In contrast to the mechanism of hGH stimulation by ghrelin, the investigators hypothesize that the supplement suppresses somatostatin, a know inhibitor of both hGH and TSH. To test this hypothesis, the investigators measured triiodothyronine (T3) after administration of the amino acid-base supplement.

DETAILED DESCRIPTION:
Two molecular targets that regulate the synthesis and secretion of human growth hormone (hGH) include 1) ghrelin, an endogenous ligand secreted by the stomach that also has appetite-stimulation properties distinct from its hGH-stimulating effects, and 2) somatostatin, a family of 14 and 28 amino acid peptides that act as a potent noncompetitive inhibitor of the release of hGH. the investigators recently reported that oral administration of a 2.9g/dose of SeroVital, a blend of l-lysine HCl, l-arginine HCL, oxo-proline, N-acetyl-l-cysteine, l-glutamine, and schizonepeta (aerial parts) powder, leads to a significant 682% mean increase in endogenous hGH levels in male and female subjects in a period of 120 minutes following acute consumption. In the work presented here, the investigators seek to characterize the mechanistic target associated with this measured increase in endogenous hGH by SeroVital, which the investigators hypothesize to be somatostatin. The investigators test this hypothesis by assaying thyroid function, a secondary inhibition target of somatostatin. The investigators further compare our findings to ghrelin-based hGH secretagogues.

ELIGIBILITY:
Inclusion Criteria:

* 12 healthy males and 4 healthy females
* Between 18 and 70 years

Exclusion Criteria:

* Pregnant or nursing
* Taking any chronic medication including birth control pills.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, M.D., Principal Investigator — Pennington Biomedical Research Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heaton AL, Kelly C, Rood J, Tam CS, Greenway FL. Mechanism for the Increase in Human Growth Hormone with Administration of a Novel Test Supplement and Results Indicating Improved Physical Fitness and Sleep Efficiency. J Med Food. 2021 Jun;24(6):653-659. doi: 10.1089/jmf.2020.0109. Epub 2020 Oct 8. PMID 33030391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were Volunteers at Pennington Biomedical Research Center, Baton Rouge, LA USA, between October 2011 and March 2011.
Pre-assignment Details: 16 participants recruited; 16 Screened, 0 excluded (12 Males and 4 Females)
Groups:
- Amino Acid Supplement First, Then Placebo: An orally administered amino acid supplement first, and after washout period, placebo.
  Placebo: A non-active orally administered supplement of the proprietary amino acid derivative
  Amino acid supplement: Supplements with the proprietary amino acid derivative blend.
- Placebo First, Then Amino Acid Supplement: Non-active Placebo first, and after washout period, an orally administered amino acid supplement.
  Placebo: A non-active orally administered supplement of the proprietary amino acid derivative
  Amino acid supplement: Supplements with the proprietary amino acid derivative blend.
Period: First Intervention
Arm/Group | Amino Acid Supplement First, Then Placebo | Placebo First, Then Amino Acid Supplement
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Wash Out Period 1 Week
Arm/Group | Amino Acid Supplement First, Then Placebo | Placebo First, Then Amino Acid Supplement
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Amino Acid Supplement First, Then Placebo | Placebo First, Then Amino Acid Supplement
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Supplements with the proprietary amino acid derivative blend.
  Amino acid supplement: An orally administered supplement of the proprietary amino acid derivative
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Triiodthyronine Over Baseline
Description: Measure Triiodthyronine at times 0-120 minutes on two occasions about one week apart. On one occasion, the proprietary amino acid derivative blend will be given orally at time 0 in capsule form, and on the other occasion the capsules will contain no amino acids.
Time Frame: 0-120 minutes, at Baseline and post dose, week 1 and week 3
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Amino Acid Supplement: Supplements with the proprietary amino acid derivative blend.
  Amino acid supplement: An orally administered supplement of the proprietary amino acid derivative
- Placebo: Non-active
  Placebo: A non-active orally administered supplement of the proprietary amino acid derivative
Arm/Group | Amino Acid Supplement | Placebo
Number analyzed (Participants) | 16 | 16
percent change | -3.3 (10.3) | -6.1 (8.5)

ADVERSE EVENTS:
Arm/Group | Amino Acid Supplement | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amino Acid Supplement (N=16) | Placebo (N=16)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No